CLINICAL TRIAL: NCT06783764
Title: Comparative Study Between Combined Modified Pectoral Nerve Block (PECSΙΙ) and Transversus Thoracic Plane Block Versus Erector Spinae Plane Block for Post-operative Analgesia Following Breast Surgeries, (randomized Clinical Trial Study)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MS560/2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Analgesia; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PECS II block and TTPB group (Active Comparator): will receive a combination of PECS II block and TTPB (injection of 10 ml 0.25% bupivacaine between pectoralis major and minor muscles and 10 ml between the pectoralis minor and serratus anterior muscles) at the third or the fourth rib, then 10 ml between the internal inter-costal muscles and the transversus thoracic muscle
  Interventions: Procedure: PECS II block and transverse thoracic plane block; Drug: bupivacaine 0.25 % injection
- ESPB group (Active Comparator): : ESPB (30 ml of 0.25% bupivacaine injected deep to the erector spinae muscle at the transverse process of the fifth thoracic vertebrae)
  Interventions: Procedure: Erector Spinae Plane Block; Drug: bupivacaine 0.25 % injection

INTERVENTIONS:
Procedure: PECS II block and transverse thoracic plane block — will receive a combination of PECS II block and TTPB (injection of 10 ml 0.25% bupivacaine between pectoralis major and minor muscles and 10 ml between the pectoralis minor and serratus anterior muscles) at the third or the fourth rib, then 10 ml between the internal inter-costal muscles and the transversus thoracic muscle
  Arms: PECS II block and TTPB group
Procedure: Erector Spinae Plane Block — ESPB (30 ml of 0.25% bupivacaine injected deep to the erector spinae muscle at the transverse process of the fifth thoracic vertebrae)
  Arms: ESPB group
Drug: bupivacaine 0.25 % injection — injection of 10 ml 0.25% bupivacaine between pectoralis major and minor muscles and 10 ml between the pectoralis minor and serratus anterior muscles) at the third or the fourth rib, then 10 ml between the internal inter-costal muscles and the transversus thoracic muscle
  Arms: PECS II block and TTPB group
Drug: bupivacaine 0.25 % injection — 30 ml of 0.25% bupivacaine injected deep to the erector spinae muscle at the transverse process of the fifth thoracic vertebrae
  Arms: ESPB group

SUMMARY:
The aim of this study is to compare the analgesic effect and safety of Modified Pectoral Nerve Block and Transverse thoracic plane block versus Erector Supine plane Block in cases undergoing modified radical mastectomy (MRM).

DETAILED DESCRIPTION:
The aim of this study is to compare the analgesic effect and safety of Modified Pectoral Nerve Block and Transverse thoracic plane block versus Erector Supine plane Block in cases undergoing modified radical mastectomy (MRM).

Primary outcome: The Nalbuphine consumption in the first 24 hours post-operative.

Secondary outcome Severity of pain will be recorded through the Visual Analogue Scale (VAS) on arrival to PACU (T0) then at 4, 8, 12, 16, 20, and 24hr postoperatively.

• Study Population: Adult female patients,aged 25-65 years undergoing modified radical mastectomy will be assigned into two equal groups using simple randomization computer generated method.

* Group A: will receive a combination of PECS II block and TTPB (injection of 10 ml 0.25% bupivacaine between pectoralis major and minor muscles and 10 ml between the pectoralis minor and serratus anterior muscles) at the third or the fourth rib, then 10 ml between the internal inter-costal muscles and the transversus thoracic muscle (Abedalmohsen, 2023).
* Group B: ESPB (30 ml of 0.25% bupivacaine injected deep to the erector spinae muscle at the transverse process of the fifth thoracic vertebrae). (Abedalmohsen, 2023).
* There's no control group.

Inclusion Criteria:

* Age 25-65 years.
* BMI 18-35.
* American Society of Anesthesiologists(ASA) Physical Status Class-I, II and III.
* Scheduled for breastsurgery.

Exclusion Criteria:

* Refusal to give written informed consent.
* History of allergy to the medications used in the study.
* Contraindications to regional anesthesia (including coagulopathy -INR>1.6, PLT<50 × 10^3/cmm- and local infection).
* Psychiatric disorder that leading to inability to cooperate, speak or read.
* BMI more than 35.
* Patients on medications for chronic pain.
* Previous anterior chest wall surgery.

Sampling Method:

Simple randomization computer guaranteed. Patients will be divided into 2 groups via sealed envelopes randomly distributed to them and will be enrolled into group A, group B.

-Sample Size: After reviewing previous study results (Abedalmohsen and Bakri, 2024) showing that among patients underwent modified radical mastectomy, the morphine consumption (mg) in postoperative follow up period was lower in patients received erector spinae plane block than in patients received erector spinae plane block (0.93 + 0.63 versus 2.13 + 0.42 respectively); a sample size of at least 40 adult female patients undergoing modified radical mastectomy divided randomly into 2 groups (20 patients in each group) will achieve 100% power, at significance level 0.05, by using Power Analysis and Sample Size Software (PASS 15) (Version 15.0.10) for sample size calculation.

Preoperative settings:

After history taking and clinical examination, routine preoperative investigations will be done to all patients including:

* Laboratory investigations as (complete blood picture, bleeding time, prothrombin time, partial thromboplastin time, Kidney function, Liver functions and viral markers)
* Imaging investigations as plain chest x-ray.
* Vas score will be explained to details to the patient and full understanding will be confirmed

Intraoperative settings:

* General anaesthesia will be carried out as per our institution protocol
* Intraoperative monitoring of ECG, HR, NIBP, SpO2 and capnography will be continued throughout the operation (Bakeer et al., 2020).

After completion of surgery and before extubation:

Group A:

All blocks will be performed by an experienced anesthetist.

US-guided PECSII block will be done on the same side of surgery with the patient lying in the supine position and the ipsilateral arm will be abducted and externally rotated, and the elbow flexed 90°.(Sonosite turbo M, Bothell, Washington, USA) and linear ultrasound probe(2.5-7.5MHZ) Transduser will be put in the ipsilateral para median sagittal plane in order to identify the coracoid process. Then the transducer is rotated slightly to allow an in-plane needle trajectory from the proximal and medial side toward the lateral side (ie, the caudal border of the transducer is moved laterally, while the proximal border remains unchanged). This rotation helps image the pectoral branch of the thoracoacromial artery.

After identification of the Pectoralis major muscle, Pectoralis minor muscle, Serratus anterior muscle and the planes in between, the 1st injection will be in the plane between the Pectoralis minor muscle and the serratus anterior muscle. The needle (disposable spinal needle, K-3 point type LUER-Lock HUB 22G) will be advanced in an in-plane technique. Two mL of normal saline will be injected to confirm the location, produce hydro-dissection, and improve needle visualization. Afterward, 20 mL of bupivacaine, 0.25%, will be injected. During the withdrawal of the needle a 2nd injection will be done in the plane between the Pectoralis major muscle and the Pectoralis minor muscle. 2ml of normal saline will be injected to produce hydro-dissection and confirm the location. 10ml of Bupivicaine 0.25% will be injected (Bakeer et al., 2020).The TTPB, 10 ml bupivacaine 0.25% was injected between the deep transversus thoracic and the superficial internal inter-costal muscles para-sternal between the third and fourth left ribs under US guidance (Abedalmohsen, 2023).

GroupB:

The ESP block will be performed positioning the patient in the lateral decubitus position with probe placement in cranio cephalad orientation by identifying the spinous process in the upper thoracic area and subsequently transverse process by moving the probe laterally as an oval hyperechoic sonographic structure. In total, 20 ml of 0.25% bupivacaine will be deposited between the erector spinae muscle and transverse process using a Sono Plex Stim cannula (21G X 100 mm, Pajunk, Germany) with the in plane technique after hydro dissection and negative aspiration. The patient will be turned supine after block placement 1gm of paracetamol, 30mg of ketorolac and 1mg Granitryl will be given to all patients. The patient will then be transferred to recovery room for follow up.(Bakeer et al., 2020).

Postoperative settings:

In the first postoperative 24 hours, VAS score will be assessed at 0, 2 ,4, 8, 12, 16 and 24 hours postoperatively.

A dose of 5 mg Naluphin will be given if VAS score exceeded 3, to maintain a score less than 3, not to exceed 20 mg per dose. IV boluses of naluphin will be given as a rescue analgesia to maintain VAS ≤ 3,

. Paracetamol 1 gm IV infusion will be given every 8 hours and ketorolac 30 mg every 12 hours postoperatively (Stormholt et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

* Age 25-65 years.
* BMI 18-35.
* American Society of Anesthesiologists(ASA) Physical Status Class-I, II and III Scheduled for breast surgery

Exclusion Criteria:

* - Refusal to give written informed consent.
* History of allergy to the medications used in the study.
* Contraindications to regional anesthesia (including coagulopathy -INR>1.6, PLT<50 × 10^3/cmm- and local infection).
* Psychiatric disorder that leading to inability to cooperate, speak or read.
* BMI more than 35.
* Patients on medications for chronic pain.
* Previous anterior chest wall surgery.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult female patients ,aged 25-65 years undergoing modified radical mastectomy
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-05 (Estimated)

PRIMARY OUTCOMES:
The Nalbuphine consumption | The first 24 hours post-operative.
  The Nalbuphine consumption in the first 24 hours post-operative.

SECONDARY OUTCOMES:
severity of pain post operative | The first 24 hours post-operative.
  Severity of pain will be recorded through the Visual Analogue Scale (VAS) on arrival to PACU (T0) then at 4, 8, 12, 16, 20, and 24hr postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt